CLINICAL TRIAL: NCT02370940
Title: Regular Consumption of High Phytate Diet Reduces Inhibitory Effect of Phytate on Nonheme Iron Absorption in Female Subjects
Brief Title: Regular Consumption of High Phytate Reduces Inhibitory Effect of Phytate on Iron Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Collaborators: HarvestPlus (Other)
Responsible Party: Principal Investigator, Dr. Manju B. Reddy, Professor, Iowa State University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IPAAD Study
Record Dates: First submitted 2015-02-11; First posted 2015-02-25 (Estimated); Last update posted 2015-02-25 (Estimated); Status verified 2015-02

CONDITIONS: Iron Bioavailability
Keywords: Iron bioavailability; phytate; serum iron curve; hepcidin; iron status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Phytate Diet (Experimental): The high phytate diet group was required to consume a high phytate diet for 8 weeks. The high phytate foods were provided for subjects. They received whole grain ready-to-eat cereals, whole wheat pasta/spaghetti, tortillas, bagels, bread and dinner rolls, corn tortillas, brown rice, canned black beans, edamame and tofu, and were encouraged to consume generous amounts of nuts and other legume products high in phytate.
  Interventions: Other: High phytate intake
- Low Phytate Diet (Experimental): The low phytate diet group was required to consume a low phytate diet for 8 weeks. They received foods similar to those for the high phytate diet group but which were made from refined wheat and white rice, eggs and cheese, and were instructed to avoid high phytate foods.
  Interventions: Other: Low phytate intake

INTERVENTIONS:
Other: High phytate intake
  Arms: High Phytate Diet
Other: Low phytate intake
  Arms: Low Phytate Diet

SUMMARY:
The purpose of this study is to investigate whether regular consumption of phytate dampens its negative effect on nonheme iron absorption.

DETAILED DESCRIPTION:
Phytate is one of the main inhibitors of nonheme iron absorption. High phytate consumption is of concern in developing countries because of the high prevalence of iron and zinc deficiency in these countries. In this study, we investigated the effect of habitual consumption of a high phytate diet on the inhibitory effect of phytate on nonheme iron absorption. Thirty-two non-anemic female subjects with ferritin ≤ 30µg/L were randomized into two groups, after matching for ferritin concentration. Each group consumed either high or low phytate foods that were provided for 8 wk. Iron bioavailability from a high phytate test meal was measured using area under the curve (AUC) for serum iron at baseline and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Marginal iron status (Serum ferritin <30ug/L)
* BMI in the range 18.5-24.9kg/m2
* Willing to modify diet to increase or decrease phytate intake
* Willing to give multiple blood samples at beginning and end of study

Exclusion Criteria:

* Pregnant
* Lactating
* Smoker
* Anemic (hemoglobin <120 g/L)
* Has gastro-intestinal disease/condition that can affect absorption

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Area under the curve for serum iron for assessing bioavailability | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Manju B Reddy, PhD, Principal Investigator — Iowa State University

REFERENCES:
- [Derived] Armah SM, Boy E, Chen D, Candal P, Reddy MB. Regular Consumption of a High-Phytate Diet Reduces the Inhibitory Effect of Phytate on Nonheme-Iron Absorption in Women with Suboptimal Iron Stores. J Nutr. 2015 Aug;145(8):1735-9. doi: 10.3945/jn.114.209957. Epub 2015 Jun 3. PMID 26041677